CLINICAL TRIAL: NCT01332604
Title: A Phase Ib, Open Label, Dose Escalation Study of the Safety and Pharmacology of GDC-0980 in Combination With a Fluoropyrimidine, Oxaliplatin, and Bevacizumab in Patients With Advanced Solid Tumors
Brief Title: GDC-0980 in Combination With a Fluoropyrimidine, Oxaliplatin, and Bevacizumab in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PIM4945g; GO00883 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-03-31; First posted 2011-04-11 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Solid Cancers
MeSH Terms: interventions — 1-(4-((2-(2-aminopyrimidin-5-yl)-7-methyl-4-morpholinothieno(3,2-d)pyrimidin-6-yl)methyl)piperazin-1-yl)-2-hydroxypropan-1-one; Bevacizumab; Capecitabine

ARMS (2):
- A (Experimental)
  Interventions: Drug: GDC-0980; Drug: capecitabine
- B (Experimental)
  Interventions: Drug: GDC-0980; Drug: bevacizumab; Drug: mFOLFOX6

INTERVENTIONS:
Drug: GDC-0980 — Oral escalating dose
Drug: bevacizumab — Intravenous repeating dose
  Arms: B
Drug: capecitabine — Oral repeating dose
  Arms: A
Drug: mFOLFOX6 — Intravenous repeating dose
  Arms: B

SUMMARY:
This is an open-label, multicenter, Phase Ib, dose-escalation study designed to assess the safety, tolerability, and pharmacokinetics of oral GDC-0980 administered in combination with capecitabine and with mFOLFOX6 chemotherapy with bevacizumab added on at Cycle 5 in patients with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented locally advanced or metastatic solid tumors for which established therapy is ineffective, not tolerable, or does not exist
* Patients with histologically or cytologically documented locally advanced or metastatic breast cancer who have received at least one prior chemotherapy-based regimen for incurable disease (Arm A)
* Patients with histologically or cytologically documented locally advanced or metastatic CRC who have not received prior oxaliplatin-based therapy within 1 year of initiation of study treatment. (Arm B)

Exclusion Criteria:

* Prior anti-cancer therapy that fulfills the following criteria: a total of more than six courses of an alkylating agent, a total of more than four courses of carboplatin-containing chemotherapy regimens, and a total of more than two courses of nitrosoureas or mitomycin C, high-dose chemotherapy requiring stem-cell support, and irradiation to >= 25% of bone marrow-bearing areas
* Current dyspnea at rest because of complications of advanced malignancy or other disease requiring continuous oxygen therapy
* Known deficiency of dihydropyrimidine dehydrogenase (DPD)
* Bisphosphonate therapy for symptomatic hypercalcemia
* Known untreated or active central nervous system (CNS) metastases
* Pregnancy, lactation, or breastfeeding

For Arm B:

* Inadequately controlled hypertension
* Prior history of hypertensive crisis or hypertensive encephalopathy
* History of myocardial infarction or unstable angina within 6 months prior to the first dose of study treatment
* History of stroke or transient ischemic attacks within 6 months prior to the first dose of study treatment
* Significant vascular disease within 6 months prior to the first dose of study treatment
* History of hemoptysis within 1 month prior to the first dose of study treatment
* Patients with one or more pulmonary tumor masses with evidence of cavitation
* Evidence of bleeding diathesis or significant coagulopathy
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first dose of study treatment
* History of abdominal fistula, GI perforation, or intra-abdominal abscess within 6 months prior to the first dose of study treatment
* Clinical signs or symptoms of GI obstruction or requirement for parenteral hydration, parenteral nutrition, or tube feeding
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Serious, non-healing wound, active ulcer, or untreated bone fracture
* The presence of an ulcerating breast cancer tumor will not render a patient ineligible
* Proteinuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-07; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 30 days after last dose of study treatment
Incidence of dose limiting toxicities (DLTs) | Up to Day 21 for Arm A and up to Day 28 for Arm B
Nature of adverse events graded according to NCI CTCAE, v4.0 | Up to 30 days after last dose of study treatment
Nature of dose limiting toxicities (DLTs)graded according to NCI CTCAE, v4.0 | Up to 28 days
Severity of adverse events | Up to 30 days after last dose of study treatment

SECONDARY OUTCOMES:
Total exposure from Time 0 to the last measurable concentration | Up to Day 2 for Arm B and up to Day 9 for Arm A
Maximum observed plasma concentration | Up to Day 2 for Arm B and up to Day 9 for Arm A
Minimum observed plasma concentration | Up to Day 2 for Arm B and up to Day 9 for Arm A
Time to maximum observed plasma concentration | Up to Day 2 for Arm B and up to Day 9 for Arm A

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (4):
- United States (3):
  - Los Angeles, California
  - Aurora, Colorado
  - Rochester, Minnesota
- Barcelona, Barcelona, Spain